CLINICAL TRIAL: NCT04219384
Title: Critical Illness Related Cardiac Arrest (CIRCA): an Investigation of the Incidence and Outcome of Cardiac Arrest Within Intensive Care Units in the United Kingdom
Brief Title: Critical Illness Related Cardiac Arrest (CIRCA)
Acronym: CIRCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Intensive Care National Audit & Research Centre (Other)
Collaborators: North Bristol NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ICNARC/02/11/2019
Record Dates: First submitted 2019-11-21; First posted 2020-01-07 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Critical Illness
Keywords: Critical Illness Related Cardiac Arrest
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critical-illness related cardiac arrest (CIRCA): Those experiencing a critical illness-related cardiac arrest in a participating adult, general ICU

SUMMARY:
CIRCA aims to determine the incidence and outcomes of in-hospital cardiac arrest (IHCA) in UK intensive care units (ICUs) and explore associated risk factors with ICU and hospital survival and quality of survival following hospital discharge.

DETAILED DESCRIPTION:
Cardiac arrest is often categorised by location, out-of-hospital or in-hospital (IHCA), as there are important differences in population characteristics and aetiology. The National Cardiac Arrest Audit (NCAA) was established to audit resuscitation teams in response to IHCA, and collects information about patient characteristics, resuscitation processes, and patient outcomes. However, it does not audit IHCAs that are not attended by the resuscitation team.

Critically ill patients managed in ICUs are experiencing failure of one or more organs and therefore more intensive and invasive therapies are needed to support these failing organs. As a result, ICUs have higher nursing and medical staffing ratios, and monitoring is usually continuous. Moreover, the skill mix of the multidisciplinary team is geared to advanced life support. Thus, the risk of cardiac arrest occurring, the involvement (or not) of the resuscitation team, and the probability of return of spontaneous circulation are all likely to be different to other IHCAs.

Accurate data on cardiac arrests in ICU are lacking and the investigators do not know how many IHCA occur in ICU in the UK, nor is the impact of an IHCA in ICU on outcome known. In addition, it is not known if these IHCAs in ICUs represent an unavoidable consequence of critical illness or, more importantly, whether they can be predicted and/or prevented.

CIRCA is a prospective, multi-centre observational cohort study nested in the Case Mix Programme (CMP) and NCAA national clinical audits. The investigators aim to determine the incidence and outcomes of IHCA in UK ICUs and explore associated risk factors with ICU and hospital survival and quality of survival following hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old or more; and either
2. Cardiac arrest (defined as receipt of chest compressions or defibrillation) occurring while in-hospital and within intensive care (defined as either ICU, HDU or combined ICU/HDU); or
3. Family member of a patient surviving to discharge from intensive care after a cardiac arrest within ICU

Exclusion Criteria:

There are no exclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults having cardiac arrest (defined as receipt of chest compressions and/or defibrillation) after admission to an Intensive Care Unit (ICU) participating in the Case Mix Programme in a hospital participating in the National Cardiac Arrest Audit
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Incidence | Up to 12 months
  Incidence of critical illness related cardiac arrest

SECONDARY OUTCOMES:
Subsequent incidence of in-hospital cardiac arrest | Up to 12 months
  Subsequent incidence of in-hospital cardiac arrest obtained through data linkage to the National Cardiac Arrest Audit
Survival status at hospital discharge | Up to 12 months
  Survival status at hospital discharge obtained from data linkage to the Case Mix Programme
Survival status at 12 months | 12 months
  Survival status at 12 months obtained from data linkage to NHS Digital
Patient quality of life measured through EQ-5D-5L questionnaire completion at 3 months | 3 months
  Patient quality of life measured through completion of EuroQol 5 Dimension (5 level) questionnaire at 3 months following critical illness related cardiac arrest
Patient quality of life measured through EQ-5D-5L questionnaire completion at 6 months | 6 months
  Patient quality of life measured through completion of EuroQol 5 Dimension (5 level) questionnaire at 6 months following critical illness related cardiac arrest
Patient quality of life measured through EQ-5D-5L questionnaire completion at 12 months | 12 months
  Patient quality of life measured through completion of EuroQol 5 Dimension (5 level) questionnaire at 12 months following critical illness related cardiac arrest
Patient quality of life measured through IQCODE questionnaire completion at 3 months | 3 months
  Patient quality of life measured through completion of Informant Questionnaire on Cognitive Decline in the Elderly questionnaire at 3 months following critical illness related cardiac arrest
Patient quality of life measured through IQCODE questionnaire completion at 6 months | 6 months
  Patient quality of life measured through completion of Informant Questionnaire on Cognitive Decline in the Elderly questionnaire at 6 months following critical illness related cardiac arrest
Patient quality of life measured through IQCODE questionnaire completion at 12 months | 12 months
  Patient quality of life measured through completion of Informant Questionnaire on Cognitive Decline in the Elderly questionnaire at 12 months following critical illness related cardiac arrest
Family member quality of life measured through FROM-16 questionnaire completion at 3 months | 3 months
  Quality of life of family member of patients surviving critical illness related cardiac arrest measured through completion of Family Reported Outcome Measures 16 questionnaire at 3 months following patient arrest
Family member quality of life measured through FROM-16 questionnaire completion at 6 months | 6 months
  Quality of life of family member of patients surviving critical illness related cardiac arrest measured through completion of Family Reported Outcome Measures 16 questionnaire at 6 months following patient arrest
Family member quality of life measured through FROM-16 questionnaire completion at 12 months | 12 months
  Quality of life of family member of patients surviving critical illness related cardiac arrest measured through completion of Family Reported Outcome Measures 16 questionnaire at 12 months following patient arrest

CONTACTS AND LOCATIONS:
Overall Officials: Matt Thomas, MD, Principal Investigator — North Bristol NHS Trust
Locations (1):
- Intensive Care National Audit & Research Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised study dataset will be available from ICNARC on request to the Chief Investigator, subject to any necessary approvals

REFERENCES:
- [Derived] Darnell R, Broomhall J, Newell C, Gendall E, Harrison D, Rowan K, Doidge J, Mouncey P, Gould D, Thomas M. Critical Illness Related Cardiac Arrest (CIRCA): a prospective investigation of the incidence and outcome of cardiac arrest within intensive care units in the United Kingdom. Resuscitation. 2025 Dec 22:110933. doi: 10.1016/j.resuscitation.2025.110933. Online ahead of print. PMID 41443583
- [Derived] Darnell R, Newell C, Edwards J, Gendall E, Harrison D, Sprinckmoller S, Mouncey P, Gould D, Thomas M. Critical illness-related cardiac arrest: Protocol for an investigation of the incidence and outcome of cardiac arrest within intensive care units in the United Kingdom. J Intensive Care Soc. 2022 Nov;23(4):493-497. doi: 10.1177/17511437211055899. Epub 2022 Mar 13. PMID 36751345